CLINICAL TRIAL: NCT02408900
Title: A Pilot Study of Muscle Ultrasound Measures as Biomarkers of Upper Motor Neuron Function
Brief Title: Muscle Ultrasound Measures as Biomarkers of Upper Motor Neuron Function
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150106; 15-N-0106
Record Dates: First submitted 2015-04-03; First posted 2015-04-06 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-08-03

CONDITIONS: Muscle Spasticity
Keywords: Spasticity; Primary Lateral Sclerosis; Elastography; Ultrasound
MeSH Terms: conditions — Muscle Spasticity; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Primary lateral sclerosis (PLS) is a rare disease. It leads to weakness in the muscle of the arms, legs, and face. People with PLS develop muscle stiffness called spasticity. Researchers want to find a better way to measure this. They want to see if ultrasound, which uses sound waves to look at parts of the body, can measure spasticity and stiffness in muscles.

Objective:

- To see if ultrasound can detect and measure muscle spasticity in people with PLS.

Eligibility:

* People ages 18 75 who have a diagnosis of PLS and are enrolled in protocol 01-N-0145.
* Healthy volunteers ages 18 75.

Design:

* Participants with PLS will have 1 study visit. Healthy participants will have upto 5 visits. Each visit will be about 2 hours.
* Participants will have tests of muscle strength. They will be examined. They will push their arms and legs against researchers in different positions.
* Participants will have tests of muscle stiffness. Their arms and legs will be moved while they relax.
* Participants will have a muscle ultrasound test. They will lie on a table. Gel will be placed on the skin over the muscles of the arms and legs. A probe, like a microphone, will be moved over the skin. Researchers will look at several muscles.
* Participants should try to stay still during the ultrasound. It may be done several times and may be done by different examiners.

DETAILED DESCRIPTION:
Objective

Persons with corticospinal, or upper motor neuron dysfunction have increased muscle stiffness from spasticity. Spasticity is established by clinical examination, but there are few reliable objective measures of spasticity. New ultrasound techniques to measure the elastic properties of tissue represent a potential measure of spasticity. The ultrasound measures of tissue elasticity are painless and quick to perform, but their ability to detect changes resulting from spasticity is uncertain. The goal of this pilot study is to see how much ultrasound measures of muscle elasticity differ between patients with spasticity and healthy controls. Secondary objectives are to correlate muscle elasticity measures with a clinical rating scale of spasticity and to assess intra and inter-rater reliability. This is a protocol for primary lateral sclerosis (PLS) patients who are enrolled in another NIH study in which they have been diagnosed with spasticity.

Study Population

23 adult PLS patients with arm or leg spasticity currently enrolled in an NIH protocol

30 healthy adult controls with normal neurological exams.

Design

The first phase, an investigator training phase, is aimed to become familiar with the Siemens Acuson S2000 after the upgrade. The two investigators will train with 5 healthy volunteers. In the second phase inter-observer variability of the ultrasound and Ashworth scale will be assessed by having healthy volunteers and patients evaluated by the different investigators. Since spasticity does fluctuate throughout the day, subjects will be consecutively assessed for inter-observer variability and within a few hours or around the same time the following day (depending on patient availability) for intra-observer variability. Each investigator will do the Ashworth scale independent of the other. Each investigator will do the ultrasound independent of the other. In the third phase, we will assess patients and volunteers to reach the sample size that a power analysis suggested that we would need to measure differences between patients with spasticity and controls.

Outcome Measures

The primary outcome will be measuring muscle stiffness from the biceps brachii using ultrasound elastography, which will be compared between patient groups and control groups. A secondary outcome will be the correlation of muscle stiffness at rest with the modified Ashworth score for elbow flexion. Measures of muscle strength and ultrasound measures of density and thickness will be examined in an exploratory fashion. Elastography of the tibialis anterior will be examined in an exploratory fashion.

ELIGIBILITY:
* INCLUSION CRITERIA:<TAB>

Healthy Controls

* Adults between ages of 18-75; matched to the patient cohort
* No history of neurological disorder
* No use of medications that produce muscle relaxation within 1 week of study, such as baclofen, cyclobenzaprine, or tizanidine.
* Able to give informed consent

Patients

* Adults between ages of 18-75
* A clinical diagnosis of primary lateral sclerosis determined in NIH protocol 01-N-0145.
* No contractures of arms and legs
* Able to give informed consent

EXCLUSION CRITERIA:

* Mechanical limitation of elbow flexion
* Achilles tendon surgical procedures
* History of cervical radiculopathy
* History of botulinum injections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-03-25; Primary Completion 2015-08-03 (Actual); Study Completion 2015-08-03 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be measuring muscle stiffness from the biceps brachii using ultrasound elastography, which will be compared between patient groups and control groups. | 2 years

SECONDARY OUTCOMES:
A secondary outcome will be the correlation of muscle stiffness at rest with the modified Ashworth score for elbow flexion. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary Kay Floeter, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States